CLINICAL TRIAL: NCT01599871
Title: Multicenter 52 Weeks Double Blind Placebo-controlled Trial for the Assessment of Theophylline on Top of Combination Therapy in Severe COPD
Brief Title: Low-dose Theophylline as Anti-inflammatory Enhancer in Severe Chronic Obstructive Pulmonary Disease
Acronym: ASSET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Son Espases (Other)
Collaborators: Spanish Research Center for Respiratory Diseases (Other); Fundación Mutua Madrileña (Other)
Responsible Party: Principal Investigator, Borja Cosio, MD, PhD, Hospital Son Espases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1559-F-447
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Theophylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Inhaled corticosteroids and long-acting beta agonist + theophylline (Slophylline capsules 100 mg/Theo-dur Retard 100 mg b.i.d.)
  Interventions: Drug: theophylline
- Control (Placebo Comparator): inhaled corticosteroids and long-acting beta agonist + Placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: theophylline — theophylline 100 mg, twice at day
  Arms: Intervention
Other: placebo — Placebo
  Arms: Control

SUMMARY:
The main objective of the study is to determine the effects of low-dose oral theophylline added to combination treatment with long-acting β-agonist (LABA) and inhaled corticosteroid (ICS) in patients with severe Chronic Obstructive Pulmonary Disease (COPD) on the rate of exacerbations defined as increase of symptoms that requires a change of medication (antibiotics and/or systemic glucocorticoid) or hospitalisation.

DESIGN: Phase III multicenter, randomized, placebo-controlled, double blind, parallel, prospective study. Patient will be recruited during an hospitalisation due to COPD exacerbation and randomised at the time of discharge to receive theophylline 100 mg or placebo on top of combination therapy with inhaled corticosteroids and long-acting beta agonist. The rate of exacerbations will be determined every three months up to one year follow-up. Cl inic visits: every 3 months (total number of clinic visits = 4). In each of them, the following information will be obtained:

* Number/severity of exacerbations or hospitalisation since last clinic visit
* Compliance and side effects
* Blood sample
* Plasma levels of theophylline
* Sputum (induced)
* MMRC
* SGRQ
* Forced spirometry + inspiratory capacity

  - At the beginning and at the end of the study
* 6MWT
* BMI
* BODE

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Ability to understand study procedures and to comply with them for the entire length of the study.
* Any gender. No contraception is required neither pregnancy expected in the range of age
* Age > 45 years
* Smoking history > 10 pack-years (current or ex-smokers)
* Clinical diagnosis of COPD
* Presence of severe airflow obstruction on forced spirometry (FEV1/FVC < 0.7 and post-BD FEV1 < 50% of reference value) staged as GOLD III or IV
* Diagnosis of COPD exacerbation on discharge.

Exclusion Criteria:

* Presence or history of other chronic respiratory diseases (asthma, bronchiectasis, TB lesions)
* Cancer
* Heart failure
* Pregnancy, or risk of pregnancy
* Other inflammatory diseases
* Previous treatment with theophylline
* For drug studies: allergy/sensitivity to study drugs or their ingredients.
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Rate of exacerbations | 1 year
  Rate of exacerbations defined as increase of symptoms that requires a change of medication (antibiotics and/or systemic glucocorticoid) or hospitalisation.

SECONDARY OUTCOMES:
Number of hospitalisation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Borja G Cosio, MD, Principal Investigator — Hospital Son Espases
Locations (10):
- Spain (10):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife, Canary Islands
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital del Mar, Barcelona
  - Hospital de Sant Pau, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Gregorio Marañón, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Cosio BG, Shafiek H, Iglesias A, Yanez A, Cordova R, Palou A, Rodriguez-Roisin R, Peces-Barba G, Pascual S, Gea J, Sibila O, Barnes PJ, Agusti A. Oral Low-dose Theophylline on Top of Inhaled Fluticasone-Salmeterol Does Not Reduce Exacerbations in Patients With Severe COPD: A Pilot Clinical Trial. Chest. 2016 Jul;150(1):123-30. doi: 10.1016/j.chest.2016.04.011. Epub 2016 Apr 21. PMID 27107490